CLINICAL TRIAL: NCT01904383
Title: Post Marketing Surveillance on Long Term Drug Use of Trazenta® Tablets as add-on Therapy in Patients With Type 2 Diabetes Mellitus
Brief Title: PMS of Trazenta on the Long-term Use as Add-on Therapy
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 1218.147
Record Dates: First submitted 2013-07-08; First posted 2013-07-22 (Estimated); Results first posted 2019-10-02 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Trazenta
  Interventions: Drug: Trazenta

INTERVENTIONS:
Drug: Trazenta — 1 tablet of 5 mg Trazenta tablets once daily

SUMMARY:
Study to investigate the safety and efficacy of long-term daily use of Trazenta® Tablets as add-on therapy in patients with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion criteria:

Patients with type 2 diabetes mellitus who are treated with anti-diabetic drugs and have never been treated with Trazenta® Tablets (linagliptin) before enrollment will be included.

Exclusion criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 3000 patients with type 2 Diabetes Mellitus
Sampling Method: Non-Probability Sample
Enrollment: 4057 (Actual)
Dates: Start 2013-07-01 (Actual); Primary Completion 2018-10-04 (Actual); Study Completion 2018-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Multiple Locations, Japan

REFERENCES:
- [Derived] Ito T, Naito Y, Shimmoto N, Ochiai K, Hayashi N, Okamura T. Long-term safety and effectiveness of linagliptin as add-on therapy in Japanese patients with type 2 diabetes: final results of a 3-year post-marketing surveillance. Expert Opin Drug Saf. 2021 Mar;20(3):363-372. doi: 10.1080/14740338.2021.1859477. Epub 2020 Dec 27. PMID 33269625

RESULTS

PARTICIPANT FLOW:
Recruitment Details: An observational, non-randomised, non-interventional study (NIS) in participants diagnosed with type 2 diabetes mellitus (T2DM) who were treated as add-on therapy were included in the surveillance based on newly collected data under routine medical practice.
  Acronym used:
  Case report form (CRF)
Pre-assignment Details: This non-randomized, post marketing surveillance (PMS) was a prospective study using a continuous investigation system. No specific criteria (e.g., demographics, baseline characteristics, concomitant drugs in use) were defined for participant enrolment. Participants were enrolled from July 2013 to September 2015.
Groups:
- Trazenta®: Participants suffering from T2DM were orally treated with Trazenta® 5 milligram (mg) tablets once daily, for 156 weeks or until discontinuation of administration.
Period: Overall Study
Arm/Group | Trazenta®
Started (Started are registered) | 4057
Treated | 3940
Completed | 2283
Not Completed | 1774
Not completed — CRF not collected | 117
Not completed — Reason not listed | 147
Not completed — Lost to Follow-up | 674
Not completed — Lack of Efficacy | 370
Not completed — Improvement | 141
Not completed — Adverse Event | 271
Not completed — No patient visit after entry | 54

BASELINE CHARACTERISTICS:
Population: Safety set: This patient set included all patients who were dispensed Trazenta® Tablets as add-on therapy, and had at least 1 observation after treatment. The patients treated with Trazenta® Tablets as monotherapy were not included.
Arm/Group | Trazenta®
Number analyzed (Participants) | 3372
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.5 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1308
  Male | 2064
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Drug Related Adverse Events
Description: Percentage of participants with drug related adverse events.
Time Frame: From first drug administration until last drug administration, up to approximately 156 weeks.
Population: as for baseline characteristics
Measure: Number; unit: Percentage (%) of participants
Arm/Group | Trazenta®
Number analyzed (Participants) | 3372
Percentage (%) of participants | 11.39

2. Secondary Outcome: The Mean Change From Baseline to Last Observation of the Treatment Period in Haemoglobin A1c (HbA1c)
Description: The mean change from baseline to last observation of the treatment period in Haemoglobin A1c (HbA1c).
Time Frame: Baseline (before administration of treatment) and last observation of the treatment period; up to 156 weeks.
Population: Efficacy set: This patient set included all patients with Trazenta® Tablets in the safety set who had a baseline and at least one available on-treatment HbA1c value and had type 2 diabetes mellitus.
Measure: Mean (Standard Deviation); unit: Percentage (%)
Arm/Group | Trazenta®
Number analyzed (Participants) | 3029
Percentage (%) | -0.49 (1.33)

ADVERSE EVENTS:
Time Frame: For Serious adverse events (AEs) and other AEs: From first drug administration until last drug administration, up to approximately 156 weeks. For All-cause mortality: From first drug administration until end of trial, up to approximately 238 weeks.
Arm/Group | Trazenta®
All-Cause Mortality (participants affected / at risk) | 74/3372
Serious Adverse Events (participants affected / at risk) | 304/3372
Other Adverse Events (participants affected / at risk) | 184/3372
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trazenta® (N=3372)
Pneumonia bacterial (Infections and infestations) | 15
Pneumonia (Infections and infestations) | 6
Gastroenteritis (Infections and infestations) | 3
Influenza (Infections and infestations) | 3
Lung infection (Infections and infestations) | 2
Peritonitis (Infections and infestations) | 2
Sepsis (Infections and infestations) | 2
Staphylococcal sepsis (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Bronchopulmonary aspergillosis (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Enterocolitis bacterial (Infections and infestations) | 1
Gangrene (Infections and infestations) | 1
Hepatitis B (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Liver abscess (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Pneumonia pneumococcal (Infections and infestations) | 1
Pyelonephritis acute (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Streptococcal infection (Infections and infestations) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Adrenal gland cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Intraductal papillary mucinous neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anaemia (Blood and lymphatic system disorders) | 5
Nephrogenic anaemia (Blood and lymphatic system disorders) | 4
Aplastic anaemia (Blood and lymphatic system disorders) | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 1
Anaphylactic shock (Immune system disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 8
Diabetes mellitus (Metabolism and nutrition disorders) | 6
Decreased appetite (Metabolism and nutrition disorders) | 5
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 3
Marasmus (Metabolism and nutrition disorders) | 3
Hyponatraemia (Metabolism and nutrition disorders) | 1
Hypophagia (Metabolism and nutrition disorders) | 1
Depression (Psychiatric disorders) | 2
Bipolar disorder (Psychiatric disorders) | 1
Psychotic disorder due to a general medical condition (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
Cerebral infarction (Nervous system disorders) | 8
Lacunar infarction (Nervous system disorders) | 5
Cerebral haemorrhage (Nervous system disorders) | 4
Subarachnoid haemorrhage (Nervous system disorders) | 3
Brain stem haemorrhage (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 2
Thrombotic cerebral infarction (Nervous system disorders) | 2
Altered state of consciousness (Nervous system disorders) | 1
Basilar artery occlusion (Nervous system disorders) | 1
Brain stem infarction (Nervous system disorders) | 1
Carotid artery stenosis (Nervous system disorders) | 1
Cerebral artery embolism (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Cerebrovascular disorder (Nervous system disorders) | 1
Hypoglycaemic coma (Nervous system disorders) | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Parkinson's disease (Nervous system disorders) | 1
Petit mal epilepsy (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Cataract (Eye disorders) | 4
Glaucoma (Eye disorders) | 1
Retinal artery occlusion (Eye disorders) | 1
Cardiac failure (Cardiac disorders) | 14
Cardiac failure congestive (Cardiac disorders) | 8
Acute myocardial infarction (Cardiac disorders) | 6
Angina pectoris (Cardiac disorders) | 6
Cardiac failure chronic (Cardiac disorders) | 6
Myocardial infarction (Cardiac disorders) | 6
Cardiac failure acute (Cardiac disorders) | 5
Cardio-respiratory arrest (Cardiac disorders) | 4
Atrial fibrillation (Cardiac disorders) | 3
Ventricular fibrillation (Cardiac disorders) | 2
Angina unstable (Cardiac disorders) | 1
Aortic valve stenosis (Cardiac disorders) | 1
Cardiac sarcoidosis (Cardiac disorders) | 1
Cardiomyopathy alcoholic (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Sinus node dysfunction (Cardiac disorders) | 1
Stress cardiomyopathy (Cardiac disorders) | 1
Tachycardia paroxysmal (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 4
Aortic aneurysm (Vascular disorders) | 1
Arteriosclerosis (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypertensive emergency (Vascular disorders) | 1
Peripheral artery occlusion (Vascular disorders) | 1
Peripheral vascular disorder (Vascular disorders) | 1
Shock haemorrhagic (Vascular disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 8
Asthma (Respiratory, thoracic and mediastinal disorders) | 3
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Eosinophilic pneumonia chronic (Respiratory, thoracic and mediastinal disorders) | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Duodenal stenosis (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 1
Large intestine polyp (Gastrointestinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Mechanical ileus (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Oesophageal ulcer (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 1
Superior mesenteric artery syndrome (Gastrointestinal disorders) | 1
Varices oesophageal (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 3
Cholangitis acute (Hepatobiliary disorders) | 3
Cholangitis (Hepatobiliary disorders) | 2
Cholecystitis acute (Hepatobiliary disorders) | 2
Hepatic cirrhosis (Hepatobiliary disorders) | 2
Cholecystitis (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1
Pemphigoid (Skin and subcutaneous tissue disorders) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1
Rapidly progressive osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1
Diabetic nephropathy (Renal and urinary disorders) | 9
Chronic kidney disease (Renal and urinary disorders) | 7
Renal impairment (Renal and urinary disorders) | 5
Renal failure (Renal and urinary disorders) | 4
Azotaemia (Renal and urinary disorders) | 3
Acute kidney injury (Renal and urinary disorders) | 2
End stage renal disease (Renal and urinary disorders) | 1
Glomerulonephritis rapidly progressive (Renal and urinary disorders) | 1
Death (General disorders) | 6
General physical health deterioration (General disorders) | 2
Sudden death (General disorders) | 2
Chest discomfort (General disorders) | 1
Drowning (General disorders) | 1
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Blood glucose increased (Investigations) | 2
Blood potassium increased (Investigations) | 1
Carbohydrate antigen 19-9 increased (Investigations) | 1
White blood cell count increased (Investigations) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 7
Fall (Injury, poisoning and procedural complications) | 6
Subdural haematoma (Injury, poisoning and procedural complications) | 4
Ankle fracture (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Hand fracture (Injury, poisoning and procedural complications) | 1
Heat illness (Injury, poisoning and procedural complications) | 1
Injury (Injury, poisoning and procedural complications) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Shunt stenosis (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trazenta® (N=3372)
Diabetes mellitus (Metabolism and nutrition disorders) | 184

LIMITATIONS AND CAVEATS:
The study was conducted in an unblinded manner and without controls. The explanatory power of the study results was limited and the study results should be interpreted with the necessary caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2013-06-07): https://cdn.clinicaltrials.gov/large-docs/83/NCT01904383/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-12): https://cdn.clinicaltrials.gov/large-docs/83/NCT01904383/SAP_001.pdf